CLINICAL TRIAL: NCT06257485
Title: Database of Transthyretin Amyloid Cardiomyopathy Cases in a Racially and Ethnically Diverse Population in the Bronx
Brief Title: Bronx Transthyretin Amyloid Cardiomyopathy Database
Status: Active, not recruiting | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-15264
Record Dates: First submitted 2024-02-05; First posted 2024-02-14 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Transthyretin Cardiac Amyloidosis; Transthyretin Amyloid Cardiomyopathy
Keywords: transthyretin cardiac amyloidosis; transthyretin amyloid cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients referred for 99mTc-pyrophosphate Single Photon Emission Computed Tomography: Patients with suspected transthyretin cardiac amyloidosis referred for 99mTc-pyrophosphate Single Photon Emission Computed Tomography
  Interventions: Diagnostic Test: 99mTc-pyrophosphate Single Photon Emission Computed Tomography

INTERVENTIONS:
Diagnostic Test: 99mTc-pyrophosphate Single Photon Emission Computed Tomography — All patients underwent 99mTc-pyrophosphate Single Photon Emission Computed Tomography and had a baseline echocardiogram

SUMMARY:
Transthyretin amyloid cardiomyopathy (ATTR-CM) is a commonly undiagnosed and potentially fatal disease. Contemporary studies on this condition often underrepresent the female gender and diverse patient populations. This registry retrospectively evaluated patients referred for 99mTc-pyrophosphate (PYP) Single Photon Emission Computed Tomography (SPECT) between 2014 and 2023 at Montefiore-Einstein in the Bronx. The patient population is racially and ethnically diverse and with a high proportion of females. Demographic, clinical (e.g. comorbidities), laboratory, echocardiographic, hospitalization, and mortality data were collected for each patient.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients referred for PYP SPECT at Montefiore Medical Center between 2014 and 2023

Exclusion Criteria:

* Did not have a transthoracic echocardiogram in our medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients referred for PYP SPECT at Montefiore Medical Center between 2014 and 2023 who had a transthoracic echocardiogram in our medical records.
Sampling Method: Non-Probability Sample
Enrollment: 476 (Estimated)
Dates: Start 2023-09-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
ATTR-CM Diagnosis | During the index PYP scan within the study time frame parameters of the retrospective review (between 2014 and 2023)
  The number of patients who underwent a PYP SPECT scan diagnostic of ATTR-CM will be assessed and reported
Mortality | Within the study time frame parameters of the retrospective review (between 2014 and 2023)
  The number of patients who died from all-cause mortality will be tabulated and reported

SECONDARY OUTCOMES:
Heart failure hospitalizations | Within the study time frame parameters of the retrospective review (between 2014 and 2023)
  The number of patients admitted to the hospital with a primary diagnosis of heart failure will be tabulated and reported
Total Hospitalizations | Within the study time frame parameters of the retrospective review (between 2014 and 2023)
  The number of patients admitted to the hospital with any diagnosis will be tabulated and reported

CONTACTS AND LOCATIONS:
Overall Officials: Leandro Slipczuk, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Health System, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Performance of Clinical Scoring Systems in the Diagnosis of Transthyretin Amyloid Cardiomyopathy in a Diverse Patient Cohort — https://pubmed.ncbi.nlm.nih.gov/39701370/